CLINICAL TRIAL: NCT00003014
Title: Carboplatin in the Adjuvant Treatment of Stage I Seminoma: A Radomized Comparison of Single Agent Carboplatin With Radiotherapy in the Adjuvant Treatment of Stage I Seminoma of the Testis, Following Orchidectomy
Brief Title: Radiation Therapy Compared With Chemotherapy in Treating Patients With Stage I Testicular Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065594; MRC-TE19; EORTC-30982; EU-97003
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2011-03

CONDITIONS: Testicular Germ Cell Tumor
Keywords: stage I malignant testicular germ cell tumor; testicular seminoma
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma | interventions — Carboplatin; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether chemotherapy is more effective than radiation therapy for testicular cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of carboplatin with that of radiation therapy in treating patients who have stage I testicular cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare relapse rates in patients with stage I testicular seminoma treated with adjuvant radiotherapy vs carboplatin. II. Compare quality of life of patients before and after treatment with these regimens. III. Compare the acute and intermediate (1-2 year) side effects of these regimens in these patients. IV. Determine the incidence of late side effects (such as bowel dysfunction) of treatment and second malignancies in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive a single dose of carboplatin IV. Arm II: Patients undergo radiotherapy once daily, 5 days a week. Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 800 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage I seminomatous germ cell tumor of the testis categorized as either "classical" or "anaplastic"

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine less than 1.4 mg/dL Other: No concurrent or previously treated malignancy except successfully treated nonmelanoma skin cancer No medical condition or other factor that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: No more than 8 weeks since prior orchidectomy Prior inguino-pelvic or scrotal surgery allowed Must be treated with "dog-leg" field if randomized to radiotherapy If prior vasectomy, choice of fields is at the discretion of the clinician

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1998-04; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Von Der Maase, MD, Study Chair — Aarhus Universitetshospital - Aarhus Sygehus; R. T. Oliver, MD, Study Chair — St. Bartholomew's Hospital
Locations (62):
- Porto Alegre Hospital, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (4):
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
- Maria Hospital, Helsinki, Finland
- Antoni van Leeuwenhoekhuis, Amsterdam, Netherlands
- Norwegian Radium Hospital, Oslo, Norway
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- United Kingdom (53):
  - Royal United Hospital, Bath, England
  - University of Birmingham, Birmingham, England
  - Children's Hospital - Birmingham UK, Birmingham, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Royal Sussex County Hospital, Brighton, England
  - Bristol Royal Hospital for Sick Children, Bristol, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Derbyshire Children's Hospital, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Gloucester Royal NHS Trust - Glouchester Royal Hospital, Gloucester, England
  - Royal Surrey County Hospital, Guildford, England
  - Royal Free Hospital, Hampstead, London, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Cookridge Hospital, Leeds, England
  - St. James's Hospital, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - Saint Bartholomew's Hospital, London, England
  - St. Bartholomew's Hospital, London, England
  - Guy's and St. Thomas' Hospitals Trust, London, England
  - Westminster Hospital, London, England
  - University College Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Manchester Children's Hospitals (NHS Trust), Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - South Tees Acute Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Newcastle Upon Tyne Hospitals NHS Trust - Freeman Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Norfolk & Norwich Hospital, Norwich, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Portsmouth Hospitals NHS Trust, Portsmouth, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Weston Park Hospital, Sheffield, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England
  - Princess Royal Hospital, Telford, England
  - Walsall Manor Hospital, Walsall, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Infirmary, Glasgow, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Llandough Hospital, Penarth, Wales
  - Royal Preston Hospital, Preston

REFERENCES:
- [Background] Mead GM, Fossa SD, Oliver RT, Joffe JK, Huddart RA, Roberts JT, Pollock P, Gabe R, Stenning SP; MRC/EORTC seminoma trial collaborators. Randomized trials in 2466 patients with stage I seminoma: patterns of relapse and follow-up. J Natl Cancer Inst. 2011 Feb 2;103(3):241-9. doi: 10.1093/jnci/djq525. Epub 2011 Jan 6. PMID 21212385
- [Result] Oliver RT, Mason MD, Mead GM, von der Maase H, Rustin GJ, Joffe JK, de Wit R, Aass N, Graham JD, Coleman R, Kirk SJ, Stenning SP; MRC TE19 collaborators and the EORTC 30982 collaborators. Radiotherapy versus single-dose carboplatin in adjuvant treatment of stage I seminoma: a randomised trial. Lancet. 2005 Jul 23-29;366(9482):293-300. doi: 10.1016/S0140-6736(05)66984-X. PMID 16039331
- [Result] Oliver RT, Mason M, Von der Masse H, et al.: A randomised comparison of single agent carboplatin with radiotherapy in the adjuvant treatment of stage I seminoma of the testis, following orchidectomy: MRC TE19/EORTC 30982. [Abstract] J Clin Oncol 22 (Suppl 14): A-4517, 386, 2004.
- [Result] Oliver RT, Mead GM, Rustin GJ, Joffe JK, Aass N, Coleman R, Gabe R, Pollock P, Stenning SP. Randomized trial of carboplatin versus radiotherapy for stage I seminoma: mature results on relapse and contralateral testis cancer rates in MRC TE19/EORTC 30982 study (ISRCTN27163214). J Clin Oncol. 2011 Mar 10;29(8):957-62. doi: 10.1200/JCO.2009.26.4655. Epub 2011 Jan 31. PMID 21282539
- [Result] Oliver RT, Mead GM, Fogarty PJ, et al.: Radiotherapy versus carboplatin for stage I seminoma: updated analysis of the MRC/EORTC randomized trial (ISRCTN27163214). [Abstract] J Clin Oncol 26 (Suppl 15): A-1, 2008.